CLINICAL TRIAL: NCT00592462
Title: Whole Body MRI for Detection of Cancer Metastases
Brief Title: Whole Body Magnetic Resonance Imaging (MRI) for Detection of Cancer Metastases
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0539; BCTR74106 (Other: Susan Komen Foundation)
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Whole Body MRI; Magnetic Resonance Imaging; Metastases
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Whole Body MRI
  Interventions: Procedure: Whole Body MRI

INTERVENTIONS:
Procedure: Whole Body MRI — The whole body MRI will include T1-weighted and T2-weighted phase-sensitive MR imaging as well as diffusion weighted imaging of the whole body in multiple patient table stations.

SUMMARY:
The objective of this pilot study is to develop and evaluate a whole body MRI technique for detecting cancer metastases. The whole body MRI will include T1-weighted and T2-weighted phase-sensitive MR imaging as well as diffusion weighted imaging of the whole body in multiple patient table stations.

DETAILED DESCRIPTION:
Researchers would like to find out if a new whole-body MRI technique is able to find cancer metastases better than a whole-body bone scan, which is the current standard of care.

Screening Tests:

Before you can start treatment on this study, you will have "screening questions" to help the doctor decide if you are eligible to take part in this study. You will be asked to complete some questionnaires to find out if there is any reason why you would not be able to receive an MRI scan. The questionnaires will cover topics such as whether you have a pacemaker and what medications you may be taking. It should take about 10-15 minutes to complete the questionnaires.

You will also have either a bone scan or positron emission tomography / computed tomography (PET/CT) during the screening period to check if the disease has spread to your bones. A bone scan is a picture that is taken, after a radioactive substance is injected into your bloodstream, allowing your doctor to see any abnormal areas of the bone. A PET/CT scan is a type of x-ray scan that uses an injected chemical to help the doctor "see" the image more clearly. For up to 6 hours before the PET/CT scan, you must not eat or drink anything except water. A small tube will be placed in your arm, and you will receive an injection of a very small amount of a mildly radioactive sugar material into your bloodstream. The radioactive nature of this injected material allows the scanner to "see" it in certain places in your body. After the injection, you will need to rest quietly until it is time for the scan. The amount of rest time may vary, but be prepared to wait for between 45 and 90 minutes. During the scan, you will lie flat on your back on a table. The scan itself may last up to 1 hour.

Study Procedures:

If you are found to be eligible and you agree to take part in this study, you will be scanned using a whole-body MRI, with and without a "contrast agent" (a chemical substance injected in your blood stream to help the scanner "see" your blood vessels better). This will be performed after you receive the bone scan as the standard of care scan.

MRI uses a large magnet instead of x-rays to take pictures of the inside of your body. People who have metal in their bodies (pacemakers, neurostimulators, certain clips, or staples from earlier surgery) may not receive an MRI. The magnetic field used in MRI scanning may harm such people or cause problems with devices such as pacemakers.

During the MRI procedure, part or all of the body will be passed into a long, narrow tube scanner, which is open at both ends. The scanner has an intercom, which will allow you to speak to the doctors and staff during the procedure. The machine will produce a loud knocking noise. This is normal. You will be given earplugs to protect your ears. The MRI will also require a line to be inserted into one of your veins to inject the contrast agent. Healthy volunteers participating in this study will not have the contrast agent injected during the scan.

Depending on how tall you are, imaging of your entire body will be achieved by the time you have been scanned at 5 or 6 different table positions. The table you are on for the scanning will be moved without having to reposition you. All images will be taken within a total scan time of about 1 hour.

The MRI findings will be compared with the bone scan that you received before the MRI. This comparison will help researchers to find out how well the MRI was able to "see" cancer metastases.

Study Length:

After the whole-body MRI, your participation in this study will be over.

This is an investigational study. All MRI scans will be performed on a commercially available GE Signa scanner (GE Healthcare, Milwaukee, WI). All the imaging techniques used will be done according to FDA MRI safety guidelines. Up to 35 patients and 5 healthy volunteers will take part in the study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer patients with high suspicion or confirmed bone metastases.
2. Patient who have undergone a clinically indicated skeletal scintigraphy within two weeks of the MRI exam.
3. Patients who have signed their informed consent form to undergo the study.

Exclusion Criteria:

1) Contraindication to conventional MR imaging (e.g. metal implants, pace maker, etc.).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Breast cancer patients with a high suspicion or confirmed bone metastases.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2007-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Develop and evaluate a whole body MRI technique for detecting cancer metastases. | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Jingfei Ma, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org